CLINICAL TRIAL: NCT05216705
Title: Study of Exploratory Plasmatic Markers of Alcohol Withdrawal
Acronym: STEP-AW
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-67
Record Dates: First submitted 2021-11-23; First posted 2022-01-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Withdrawal
Keywords: biomarkers; alcohol use disorder; alcohol withdrawal; central nervous system; alcohol brain damage
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasmatic samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research focuses on alcohol withdrawal in hospitals and its potential neurological consequences.

Alcohol withdrawal is an event that induces physical symptoms, such as tremors, sweating, anxiety and requires medical support. Sometimes alcohol withdrawal results in neurological complications, such as epileptic seizures, delirium tremens, Wernicke Encephalopathy, memory and cognitive disorders. Chronic alcohol consumption and lack of vitamin B1 also cause neurological damage. Magnetic resonance imaging of the brain can be used to assess severe forms, but gives little information about possible recovery and mild or transient forms.

Currently, there is no scientifically validated blood measurement to assess the intensity of these neurological complications, to predict their occurrence and recovery, or to distinguish between the consequences of chronic alcohol consumption, complications of alcohol withdrawal and vitamin B1 deficiency.

This is non-experimental, non-controlled observational research.

Four plasma biomarkers were selected to be evaluated in the field of alcoholology. t is the dosage of light neurofilaments (NFL), the Tau protein, the glial fibrillary acidic protein (GFAP) and the ubiquitin carboxyl terminal hydrolase L1 (UCHL-1). These biomarkers are studied, in particular in cerebrospinal fluid, in neurodegenerative diseases and in patients having experienced a cranial trauma. They were described in the literature as markers of cerebral suffering. NF-L would reflect the axon injury, Tau and UCHL-1 protein the neurons injury and GFAP the astrocytes injury. The Quanterix* assay technique (SIMOA technology) allows simultaneous assay of these 4 biomarkers, with a detection threshold 100 times lower than that of the ELISA technique. This allows plasma assays to be performed and is therefore more accessible and less risky for the patient than assays in cerebrospinal fluid.

The objective was to study the kinetics of these four biomarkers (NFL, Tau, GFAP, UCHL-1) during alcohol withdrawal, it was decided to measure these plasma biomarkers at three points during alcohol withdrawal : at the beginning of withdrawal (T1 = J1), after the time when withdrawal is most intense and complications such as Wernicke Encephalopathy or delirium tremens usually occur (T2 = J3-J4), and at the end of alcohol withdrawal management (T3 = J13-J15).

The choice of performing T1 the day after the patient's admission (D1) and not the day of the patient's admission (D0) was determined to allow a better homogeneity of the plasma assay and to respect the reflection period before signing the consent. Indeed, patients may have different levels of alcohol in their blood when they are admitted on the morning of D0. This induces a heterogeneous clinic and interferes with the interview and the delivery of an informed information. Moreover, the dosage thus carried out at D1 will be done fasting, on waking, while the patient will be non-alcoholic, under identical conditions for all patients.

In this exploratory study, the number of subjects needed is set at 18 subjects who have completed the research, i.e., having had three samples at D1 (T1), D3-J4 (T2) and D13-J15 (T3) without alcohol consumption until T3. Subjects leaving the study before this third test will be replaced up to a maximum of 7 replacements. With no previous study to our knowledge measuring these biomarkers in alcohol withdrawal, we cannot anticipate the variance. We therefore set the number of subjects to be included based on the capacity of a SIMOA assay kit for the four biomarkers NLF, Tau, GFAP, and UCHL-1. Anticipating, the risk of alcohol reconsumption, early discharge and lost to follow-up, it is planned to include 25 patients. Inclusions will end after the third follow-up visit (T3) of the 18th patient for whom we will have all three samples taken (complete data) or after T3 of the 25th patient included.

The risks for the patient are the occurrence of a complication during the procedures included in the protocol, i.e. for all patients, one or more haematomas at the points of venous sampling or the occurrence of a vagal malaise.

ELIGIBILITY:
Inclusion Criteria:

* Admission for inpatient alcohol withdrawal (planned or unplanned)
* Last alcohol consumption less than 24 hours before admission to hospital
* Active alcohol use disorder (DSM 5 criteria)
* Age 18 to 65 years
* Affiliation to a social welfare system or beneficiary of such a system.

Exclusion Criteria:

* Active use disorder of benzodiazepines, delta-9-tetrahydrocannabinol (THC), opioids, cocaine, amphetamines, new synthetic drug, gamma-hydroxybutyrate/gamma-butyrolactone, hallucinogens, assessed by interview
* Use in the previous 30 days of THC, opioids, cocaine, amphetamines, a new synthetic product, gamma-hydroxybutyrate/gamma-butyrolactone, hallucinogenic substances, assessed by questioning or positive by urine test,
* Patient on opioid maintenance therapy (methadone or buprenorphine)
* Presence of decompensated cirrhosis (Child Pugh score B or C) on admission or liver insufficiency with a TP < 70%,
* Presence of severe acute alcoholic hepatitis (Maddrey score ≥32) on admission,
* Presence of chronic renal failure with a glomerular filtration rate of less than 60mL/minute/1.73m2 estimated by the Cockroft formula,
* Presence of acute renal failure,
* Presence of another condition that may cause brain damage :
* epileptic seizure, stroke, head trauma within the last three months,
* previously diagnosed severe cognitive impairment
* history or active infection with HIV, hepatitis C virus (HCV) or syphilis, known and noted in the medical record, collected in the history or noted in the systematic screening for sexually transmitted infections carried out for care,
* Patient with a language barrier (unable to follow the protocol or respond to clinical assessments),
* Hospitalization expected to be less than 15 days and not able to perform the protocol assay at D14,
* Pregnant, parturient or breastfeeding women,
* Person deprived of liberty by judicial or administrative decision,
* Person hospitalised without consent and not subject to a legal protection measure,
* Person subject to an exclusion period for other research,
* Adult person subject to a legal protection measure, adult person unable to express his or her consent and not subject to a protection measure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population of the study STEP-AW is the male and female patients, aged 18 to 65 years inclusive, admitted for inpatient alcohol withdrawal.
  In terms of the number of patients included, it is planned to include up to a maximum of 25 patients to obtain 18 patients with the three samples performed (i.e. 7 replacements maximum).
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Change in NFL between T1 and T3 | day 1 to day 15
  The primary endpoint of the STEP-AW study will be the change in the measurement of the biomarkers at T1 (D1 of admission for alcohol withdrawal, i.e. at the start of withdrawal) and T3 (D13-D15, i.e. once alcohol withdrawal has been completed)
Change in Tau protein between T1 and T3 | day 1 to day 15
  The primary endpoint of the STEP-AW study will be the change in the measurement of the biomarkers at T1 (D1 of admission for alcohol withdrawal, i.e. at the start of withdrawal) and T3 (D13-D15, i.e. once alcohol withdrawal has been completed)
Change in GFAP between T1 and T3 | day 1 to day 15
  The primary endpoint of the STEP-AW study will be the change in the measurement of the biomarkers at T1 (D1 of admission for alcohol withdrawal, i.e. at the start of withdrawal) and T3 (D13-D15, i.e. once alcohol withdrawal has been completed)
Change in UCHL1 between T1 and T3 | day 1 to day 15
  The primary endpoint of the STEP-AW study will be the change in the measurement of the biomarkers at T1 (D1 of admission for alcohol withdrawal, i.e. at the start of withdrawal) and T3 (D13-D15, i.e. once alcohol withdrawal has been completed)

SECONDARY OUTCOMES:
Change in biomarkers between T1 and T2 | day 1 to day 4
  Test of the difference in the measurement of these biomarkers at T1 (D1) and at T2 (D3-D4 of admission for alcohol withdrawal).
Correlation of the change between T1 and T3 of the four biomarkers | day 1 to day 15
  The correlation of the change between T1 and T3 in the levels of these four plasmatic biomarkers with each other (NFL, Tau, GFAP, UCHL-1)
Correlation with the plasmatic glutamate | day 1 to day 15
  Correlation of the change between T1 and T3 of the four biomarkers with the change of the plasmatic glutamate between T1 and T3
Association with the intensity of alcohol withdrawal | day 1 to day 15
  The association of the change between T1 and T3 in these biomarkers with the intensity of alcohol withdrawal at D1, expressed as the dose of benzodiazepine required to control withdrawal signs over the whole day of D1 (maximum daily dose during withdrawal).
Association with neurological signs | day 1 to day 15
  Association of the change between T1 and T3 of these biomarkers with signs of neurological severity of alcohol withdrawal at T1 expressed by the presence of clinical signs of the Wernicke Encephalopathy triad (ophthalmoplegia, ataxia, confusion).

CONTACTS AND LOCATIONS:
Locations (1):
- GHU APHP Nord - Université de Paris, Site Lariboisière Fernand-Widal, Paris, France